CLINICAL TRIAL: NCT01174238
Title: A Two Arm Phase II Trial of Sequential Axitinib and Carboplatin/Paclitaxel in Melanoma With Correlative FLT PET Scans (3'Deoxy-3'-18F-Fluorothymidine Positron Emission Tomography Scans)(CC# 10852)
Brief Title: A Two Arm Trial of Axitinib and Carboplatin/Paclitaxel in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adil Daud (Other)
Responsible Party: Sponsor-Investigator, Adil Daud, Clinical Professor, Hem/Onc, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10852
Record Dates: First submitted 2010-07-28; First posted 2010-08-03 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Melanoma
Keywords: Melanoma; Axitinib; Carboplatin; Paclitaxel
MeSH Terms: conditions — Melanoma | interventions — Axitinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients enrolled in Arm A and Arm B will receive the same treatment with study drugs axitinib, carboplatin, and paclitaxel. Patients enrolled in Arm A and Arm B will have tumor imaging assessments: PET-CT, CT Scan, and/or MRI. In addition patients enrolled in Arm A will also have FLT-PET scans.
  Interventions: Drug: Axitinib; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (Experimental): Patients enrolled in Arm A and Arm B will receive the same treatment with study drugs axitinib, carboplatin, and paclitaxel. Patients enrolled in Arm A and Arm B will have tumor imaging assessments: PET-CT, CT Scan, and/or MRI. Patients enrolled in Arm B will not have FLT-PET scans.
  Interventions: Drug: Axitinib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Axitinib — 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
Drug: Carboplatin — Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
Drug: Paclitaxel — Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.

SUMMARY:
This is a two arm prospective Phase II pilot trial designed to determine the optimal duration of break between axitinib and chemotherapy with carboplatin/paclitaxel in melanoma. In this study, 6 patients will be enrolled to Arm A, the FLT PET scan (3'deoxy-3'-18F-Fluorothymidine positron emission tomography scans)cohort. 30 patients will be enrolled to Arm B, the treatment-only cohort. 36 total patients will be enrolled. The treatment schedule will be the same in either cohort, with the exception of the FLT PET scans.

DETAILED DESCRIPTION:
This is a two arm prospective Phase II pilot trial designed to determine the optimal duration of break between axitinib and chemotherapy with carboplatin/paclitaxel in melanoma. In this study, 6 patients will be enrolled to Arm A, the FLT-PET (3'deoxy-3'-18F-Fluorothymidine positron emission tomography scans)cohort. 30 patients will be enrolled to Arm B, the treatment-only cohort. 36 total patients will be enrolled. The treatment schedule and dose will be the same in either cohort, with the exception of the FLT PET scans. We are enrolling only 6 patients to Arm A, the FLT-PET cohort, because of study financial considerations.

Patients will be enrolled in Arm A first, the FLT-PET cohort, to accommodate the radiological manufacture of the FLT-PET scan dye. It is expensive to manufacture and it is not usable forever. However if a patient is unable to participate in Arm A because of logistical issues, i.e. not being able to travel to UCSF for FLT-PET scans we will offer them participation in Arm B so that they can receive treatment that is not available off study.

Each treatment cycle will last for 21days. During Cycle 1, patients will be treated with:

Days 1-14: axitinib 5 mg PO twice daily Days 15-21: break from treatment

In all cycles after Cycle 1, patients will be treated with:

Day 1: paclitaxel 175 mg/m2 over 3 hours followed by carboplatin AUC 5 (AUC 5 is a term used to describe the dosing of carboplatin based on a patient's height, weight and kidney function) over 45 minutes Days 1-14: axitinib 5 mg PO twice daily Days 15-21: break from treatment Arm A: FLT PET cohort subjects will have FLT PET scans up to 2 weeks prior to day 1 and on days 14, 17, and 21 of cycle 1.

Arm B: Treatment-only patients will receive administration of axitinib and carboplatin/paclitaxel on the same schedule and dose as Arm A but will not have FLT PET scans. Patients in Arm B will have standard tumor assessment with FDG PET-CT scans (F18-deoxyglucose positron emission tomography scans), CT Scans, and MRI's.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven melanoma with Stage IV or unresectable stage III disease.
2. Male or female, age ≥ 18 years.
3. Resolution of all acute toxic effects of prior radiotherapy, chemotherapy or surgical procedures to NCI CTCAE Version 4.0 grade ≤1.
4. May have ≤ 2 prior chemotherapy treatments and any prior immunotherapy treatments. These can include dacarbazine and/or temozolomide but not carboplatin or paclitaxel.
5. At least 2 weeks since the end of prior systemic treatment (4 weeks for bevacizumab-containing regimens), radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤ 1 or back to baseline except for alopecia or hypothyroidism.
6. No evidence of preexisting uncontrolled hypertension. The baseline systolic blood pressure readings must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
7. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   2. Total serum bilirubin ≤ 1.5 x ULN (Grade 0-1)
   3. Absolute neutrophil count (ANC) ≥ 1500 /ml
   4. Platelets ≥ 100,000/mL
   5. Hemoglobin ≥ 9.0 g/dL (may be transfused or erythropoietin treated)
   6. Serum calcium ≥12.0 mg/dL
   7. Serum creatinine ≤ 1.5 x ULN
8. Patients with CNS (central nervous system) metastasis must have had either:

   1. Resected CNS metastasis without evidence of recurrence for > 12 weeks, OR
   2. Brain metastasis treated by stereotactic radiosurgery without evidence of recurrence or progression for 12 weeks, OR
   3. Multiple brain lesions treated with whole brain radiation therapy with stable disease off corticosteroids for at least 12 weeks prior to the start of therapy, AND
   4. Without any evidence of leptomeningeal disease, AND
   5. Patients must be neurologically intact.
9. May have previous adjuvant therapy with interferon, vaccines, or therapy with IL-2 or GM-CSF.
10. Measurable disease by RECIST criteria.
11. ECOG performance status 0 or 1.

Exclusion Criteria:

1. Major surgery within 4 weeks of starting the study treatment.
2. Radiation therapy within 2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
3. NCI CTCAE version 4.0 grade 2 or greater hemorrhage within 4 weeks of starting study treatment.
4. History of hemoptysis or bleeding from GI tract.
5. History of abdominal fistulae or perforation within 6 months prior to starting study treatment.
6. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease on screening CT or MRI scan.
7. Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
8. Hypertension that cannot be controlled by medications.
9. Current use or anticipated need for treatment with drugs that are known potent CYP3A inhibitors (grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine).
10. Current use or anticipated need for treatment with drugs that are known potent CYP3A or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
11. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
12. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
13. CNS disease on stable dexamethasone
14. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
15. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, MD, Principal Investigator — Cutaneous Oncology Group at the Helen Dillar Family Comprehensive Cancer Center at UCSF
Locations (1):
- Cutaneous Onocology Group at the Helen Dillar Family Comprehensive Cancer Center UCSF, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients were consented; two participants were lost to follow-up prior to treatment and hence were not included in any analyses
Groups:
- Axitinib + Carboplatin/Paclitaxel: Axitinib: 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
  Carboplatin: Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.
Period: Overall Study
Arm/Group | Axitinib + Carboplatin/Paclitaxel
Started | 38
Participants That Underwent FLT-PET Scan | 6
Completed | 36
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: of 40 consented participants, 38 received at least one study treatment
Groups:
- Axitinib+Carboplatin/Paclitaxel, Including FLT-PET Patients: Axitinib: 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
  Carboplatin: Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.
  6 patients in this group received drug treatment and in addition underwent FLT-PET during first treatment cycle.
Arm/Group | Axitinib+Carboplatin/Paclitaxel, Including FLT-PET Patients
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients with tumor size reduction, i.e. the sum of partial responses plus complete responses. Radiographic response was evaluated using RECIST criteria during every 21-day cycle of treatment.
Time Frame: Monthly during study treatment, up to 12 months
Population: Two patients discontinued treatment due to toxicity within the first 3 weeks, prior to the first infusion of paclitaxel/carboplatin, and were considered to be evaluable for toxicity but not for response.
Measure: Number; unit: percentage of patients
Groups:
- Axitinib + Carboplatin/Paclitaxel: All enrolled patients received the same treatment with study drugs axitinib, carboplatin, and paclitaxel and had tumor imaging assessments: PET-CT, CT Scan, and/or MRI. 6 of 38 patients were selected to undergo FLT-PET scans.
  1 treatment cycle: 21 days
  * dual therapy: 5mg Axitinib on days 1-14, twice a day (BID)
  * monotherapy: if patient completes ≥ 6 cycles, 5mg Axitinib every day, once a day (QD)
  Carboplatin: Day 1 of each treatment cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients in dual therapy phase.
Arm/Group | Axitinib + Carboplatin/Paclitaxel
Number analyzed (Participants) | 36
percentage of patients | 22

2. Secondary Outcome: Optimal Interval Between the End of Axitinib Therapy and Initiation of Chemotherapy
Description: Optimal interval between the end of axitinib therapy and initiation of chemotherapy, as determined using FLT PET as a Radiological Biomarker information of Resumption of DNA Synthesis Following Axitinib Therapy.
Time Frame: Days 1, 14, 17, and 20 of cycle 1
Measure: Number; unit: days
Groups:
- Axitinib + Carboplatin/Paclitaxel With FLT-PET Scans: Axitinib: 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
  Carboplatin: Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.
Arm/Group | Axitinib + Carboplatin/Paclitaxel With FLT-PET Scans
Number analyzed (Participants) | 5
days | 7

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the duration from first dose of study medication to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline until death or up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Axitinib+Carboplatin/Paclitaxel, Including FLT-PET Patients: Axitinib: 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
  Carboplatin: Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.
  6 patients underwent FLT-PET during first treatment cycle.
Arm/Group | Axitinib+Carboplatin/Paclitaxel, Including FLT-PET Patients
Number analyzed (Participants) | 36
months | 14.0 [10.0 to 17.9]

4. Secondary Outcome: Time to Progression (TTP)
Time Frame: within 7 days of odd cycles after cycle 1 for the duration of treatment, up to 12 cycles
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib+Carboplatin/Paclitaxel, Including FLT-PET Patients
Number analyzed (Participants) | 36
months | 8.7 [5.5 to 12.0]

5. Secondary Outcome: Increase From Nadir in the Sum of Maximum (18)F-FLT Uptake Values After Treatment Holiday
Description: (18)F-FLT uptake values following a 7-day treatment holiday compared to the lower of Baseline or Day 14 value.
Time Frame: Baseline, Day 14, Day 20
Population: Five patients completed both pre- and post-treatment (18)F-FLT PET scans; one patient had minimal (18)F-FLT uptake at baseline
Measure: Number; unit: participants
Arm/Group | Axitinib + Carboplatin/Paclitaxel With FLT-PET Scans
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: Patients were assessed during study treatment for adverse events up to 12 months
Groups:
- Axitinib + Carboplatin/Paclitaxel and With FLT-PET Scans: Axitinib: 5mg BID Axitinib Days 1-14 for dual therapy - 5mg BID QD for patients on monotherapy
  Carboplatin: Day 1 of each 21 day cycle in combination with paclitaxel if patients are in dual therapy phase
  Paclitaxel: Day 1 of each 21 Day cycle in combination with Carboplatin if patients on on dual therapy phase.
  FLT-PET during first treatment cycle.
Arm/Group | Axitinib + Carboplatin/Paclitaxel | Axitinib + Carboplatin/Paclitaxel and With FLT-PET Scans
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/6
Serious Adverse Events (participants affected / at risk) | 12/32 | 1/6
Other Adverse Events (participants affected / at risk) | 32/32 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Carboplatin/Paclitaxel (N=32) | Axitinib + Carboplatin/Paclitaxel and With FLT-PET Scans (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Other (Infections and infestations) | 2 | 1
Appendicitis (Surgical and medical procedures) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
anorexia (Metabolism and nutrition disorders) | 2 | 0
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
confusion (Nervous system disorders) | 2 | 0
acute kidney disease (Renal and urinary disorders) | 1 | 0
anemaia (Blood and lymphatic system disorders) | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
thromboembolic event (Vascular disorders) | 1 | 0
heart failure (Cardiac disorders) | 1 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
other (Psychiatric disorders) | 1 | 0
transient ischemic attack (Vascular disorders) | 2 | 0
ataxia (Nervous system disorders) | 1 | 0
dizziness (Blood and lymphatic system disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 2 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0
urinary tract infection (Infections and infestations) | 1 | 0
failure to thrive (General disorders) | 1 | 0
fever (Infections and infestations) | 1 | 0
chest pain (Cardiac disorders) | 1 | 0
supraventricular tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Carboplatin/Paclitaxel (N=32) | Axitinib + Carboplatin/Paclitaxel and With FLT-PET Scans (N=6)
Fatigue (General disorders) | 27 | 5
Chills (General disorders) | 7 | 1
Gait disturbance (General disorders) | 4 | 2
Edema limbs (General disorders) | 5 | 0
Non-cardiac chest pain (General disorders) | 5 | 0
Pain (General disorders) | 5 | 0
Fever (General disorders) | 3 | 1
Infusion related reaction (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 21 | 4
Diarrhea (Gastrointestinal disorders) | 20 | 3
Constipation (Gastrointestinal disorders) | 18 | 4
Vomiting (Gastrointestinal disorders) | 13 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 2
Mucositis oral (Gastrointestinal disorders) | 4 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Bloating (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 5
Dizziness (Nervous system disorders) | 12 | 4
Headache (Nervous system disorders) | 9 | 3
Dysgeusia (Nervous system disorders) | 7 | 2
Paresthesia (Nervous system disorders) | 4 | 2
Memory impairment (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 3 | 0
Ataxia (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 2 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 2
Transient ischemic attacks (Nervous system disorders) | 2 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Spasticity (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 15 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 14 | 4
Hypotension (Vascular disorders) | 2 | 2
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 10 | 2
Platelet count decreased (Investigations) | 10 | 2
Weight loss (Investigations) | 6 | 1
Investigations - Other, specify (Investigations) | 3 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 3
Confusion (Psychiatric disorders) | 5 | 1
Depression (Psychiatric disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Blurred vision (Eye disorders) | 10 | 2
Eye disorders - Other, specify (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 4 | 1
Appendicitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hypothyroidism (Endocrine disorders) | 7 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 4 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 3
Urinary urgency (Renal and urinary disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes